CLINICAL TRIAL: NCT01615367
Title: Nutrition, Exercise, and Wellness Treatment (NEW Tx) for Bipolar Disorder
Acronym: NEW Tx
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Instructor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH091182-02 (NIH)
Record Dates: First submitted 2012-05-31; First posted 2012-06-08 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Nutrition; Exercise; Symptoms; Functioning
MeSH Terms: conditions — Bipolar Disorder; Motor Activity | interventions — Nutritional Status; Exercise; Health; Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NEW Tx (Experimental): 25 people will be randomized to NEW Tx, a weekly individualized psychotherapy. Therapy is 20 weeks long.
  Interventions: Other: Nutrition, Exercise, and Wellness (NEW) psychotherapy
- Treatment as usual (TAU) (Active Comparator): 25 people will be randomized to TAU and will meet with their psychiatrist as often as clinically needed over the 20 week study duration.
  Interventions: Drug: Typically consists of at least one FDA-approved mood stabilizer

INTERVENTIONS:
Other: Nutrition, Exercise, and Wellness (NEW) psychotherapy — NEW Tx is a flexible modular treatment such that modules are selected based on the needs of the individual to increase its generalizability across patients, settings, and providers as well as its acceptability to patients.
  Arms: NEW Tx
Drug: Typically consists of at least one FDA-approved mood stabilizer — Pharmacotherapy will be conducted by experts in BD treatment and will follow the empirically-supported treatment algorithm for BD that has been developed and recently revised. The foundation of TAU is to maintain treatment with at least one Food and Drug Administration approved mood stabilizer. For TAU, medication and dosage changes are allowed as needed as long as the change is recommended based on the guidelines and participants remain on a mood stabilizer.
  Arms: Treatment as usual (TAU)

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in bipolar disorder, yet no empirically validated psychosocial interventions to manage risk factors for CVD in BD have been developed. The purpose of this study is to develop and test the feasibility of an integrated treatment to decrease CVD risk factors, while exploring whether the intervention improves overall functioning and mood symptoms. The designed treatment integrates theories on Nutrition strategies, Exercise interventions, and Wellness Treatment (NEW Tx) to address risk factors for CVD that co-occur with bipolar disorder. NEW Tx includes novel intervention strategies in each of these three modules, as well as modified and tailored empirically-supported strategies for bipolar disorder. The primary hypotheses are that NEW Tx will be feasible to deliver, acceptable to this population, and associated with improvements in CVD risk factors (i.e., waist circumference). Exploratory analyses will examine predictors of treatment response and the effect of NEW Tx on mood symptoms and overall functioning.

DETAILED DESCRIPTION:
The purpose of the Nutrition, Exercise, and Wellness Treatment (NEW Tx) research is to develop and test the feasibility and acceptance of a theoretically integrated treatment to address the impact of medical comorbidity of individuals with bipolar disorder (BD), while exploring its efficacy, whether it improves overall functioning and symptoms, as well as examine a potential moderator and mediator of treatment response.

A.Primary Aims

Aim 1: Feasibility and Acceptance of NEW Tx in the Nonrandomized Trial.

Hypothesis 1a: A preliminary study of whether NEW Tx will be feasible with regards to recruitment, retention, blinded assessments, and therapist adherence to NEW Tx.

Hypothesis 1b: Participants will report high satisfaction with the treatment and acceptability over the study duration in a nonrandomized trial.

Aim 2: Feasibility and Acceptance of NEW Tx and its Evaluation in the Randomized Pilot Trial.

Hypothesis 2a: A pilot study of whether NEW Tx will be feasible with regards to recruitment, randomization, retention, blinded assessments, and therapist adherence to NEW Tx.

Hypothesis 2b: Participants will report high satisfaction with the treatment and acceptability over the study duration in the randomized pilot trial.

B. Exploratory Aims

Aim 3a: Reducing Medical Burden in the Randomized Pilot Trial. Pilot test the efficacy of NEW Tx in improving medical burden using the Framingham Risk Score (FRS).

Hypothesis 3a: Over the course of 20-weeks (18 sessions) the NEW Tx group will have a lower FRS compared to treatment as usual (TAU) in the randomized pilot trial.

Aim 3b: Symptoms and Functioning in the Randomized Pilot Trial. Examine the efficacy of NEW Tx in improving functioning and symptoms of BD.

Hypothesis 3b: Over the course of 20-weeks (18 sessions) the NEW Tx group will improved functioning and mood symptoms compared to TAU in the randomized pilot trial.

Aim 3c: Moderator and Mediator of NEW Tx in the Randomized Pilot Trial. Investigate a potential moderator and mediator of treatment response.

Hypothesis 3c.1: Individuals with higher baseline Body Mass Index (BMI) > 30 will moderate the between treatment effect size for medical burden (FRS) in the randomized pilot trial, such that of NEW Tx will have lower FRSs.

Hypothesis 3c.2: Mastery of the diet and exercise modules of NEW Tx will mediate the association of NEW Tx and improvement in medical burden (FRS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder (Type I or II), which is the primary focus of treatment
* Ability to give informed consent
* Currently ill (CGI-BP ≥ 3)
* Age > 18 years and < 65 years
* Overweight individuals (BMI > 25)

Exclusion Criteria:

* Unwilling/unable to comply with study procedures
* Endorsed item, confirmed by patient's physician, on the PAR-Q
* Euthymic (CGI-BP < 3)
* Diagnosis of an eating disorder (e.g., anorexia nervosa, bulimia nervosa) in the past month
* Diagnosis of substance dependence in the past month
* Active suicidality (MADRS item 9 score > 4)
* Pregnant (as analyzed by a urine pregnancy test)
* Currently receiving another psychosocial treatment
* Exercising regularly (i.e., 5 days per week for 30 min)
* Neurologic disorder or history of head trauma
* Contraindications to exercise or diet interventions (e.g., co-morbid nutritional and metabolic diseases, physical injuries)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NEW Tx: 19 people were randomized to NEW Tx, a weekly individualized psychotherapy. Therapy is 20 weeks long.
  Nutrition, Exercise, and Wellness (NEW) psychotherapy: NEW Tx is a flexible modular treatment such that modules are selected based on the needs of the individual to increase its generalizability across patients, settings, and providers as well as its acceptability to patients.
- Treatment as Usual (TAU): 19 people were randomized to TAU and will meet with their psychiatrist as often as clinically needed over the 20 week study duration.
  Typically consists of at least one FDA-approved mood stabilizer: Pharmacotherapy will be conducted by experts in BD treatment and will follow the empirically-supported treatment algorithm for BD that has been developed and recently revised. The foundation of TAU is to maintain treatment with at least one Food and Drug Administration approved mood stabilizer. For TAU, medication and dosage changes are allowed as needed as long as the change is recommended based on the guidelines and participants remain on a mood stabilizer.
  Participants randomized to TAU who complete the first 20 weeks of the study will have the option to receive NEW Tx. TAU participants who chose to receive NEW Tx (the waitlist group) will follow the same procedures as the NEW Tx group over an additional 20 weeks. Assessment data was collected but not analyzed.
Period: Overall Study
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Started | 19 | 19
Completed | 14 | 13 (11 TAU participants chose to participate in NEW Tx after the completion of the waitlist period.)
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual (TAU): 19 people were randomized to TAU and will meet with their psychiatrist as often as clinically needed over the 20 week study duration.
  Typically consists of at least one FDA-approved mood stabilizer: Pharmacotherapy will be conducted by experts in BD treatment and will follow the empirically-supported treatment algorithm for BD that has been developed and recently revised. The foundation of TAU is to maintain treatment with at least one Food and Drug Administration approved mood stabilizer. For TAU, medication and dosage changes are allowed as needed as long as the change is recommended based on the guidelines and participants remain on a mood stabilizer.
- Total: Total of all reporting groups
Arm/Group | NEW Tx | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index level at baseline.
  kg/m^2 | 33.99 (4.47) | 36.37 (6.75) | 35.18 (5.78)
Weekly Exercise Duration [Mean (Standard Deviation); unit: minutes] — Weekly exercise duration reported at baseline.
  minutes | 26.05 (34.50) | 65.00 (74.99) | 45.00 (60.33)
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale is a 10-item clinician-rated measure of depression that assesses the presence and severity of patient's current depressive symptoms. The score for each item is summed for a total score that ranges from 0 to 60 with higher scores indicating more severe current depressive symptoms.
  units on a scale | 13.39 (9.06) | 12.37 (9.23) | 12.86 (9.03)
Young Mania Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Young Mania Rating Scale is an 11-item, clinician-rated measure that assesses the presence and severity of patient's current symptoms of mania. The score for each item is summed for a total score that ranges from 0 to 56 with higher scores indicating more severe current manic symptoms.
  units on a scale | 5.42 (8.55) | 5.95 (5.90) | 5.68 (7.25)

OUTCOME MEASURES:

1. Primary Outcome: NEW Tx Scale
Description: NEW Tx Scale is a 10-item scale to asses participants' expectations of NEW Tx their acceptability of NEW Tx at Week 20. This scale also includes a comments section to solicit unstructured feedback from participants on NEW Tx. The scale for this item is a 5-point Likert scale ranging from 1 ("strongly agree") to 5 ("strongly disagree"). The score for each item is summed for a total score that ranges from 10 to 50 with higher scores indicating poorer perception of the treatment. TAU participants only received this questionnaire if they chose to participate in the NEW Tx at week 20 of the intervention following the waitlist period.
Time Frame: 20 weeks
Population: Participants in the treatment as usual condition were not required to complete this assessment if they did not elect to complete the NEW Tx intervention following the waitlist period. Participants completed this survey at the post-treatment visit only. Results only includes data from participants who completed the treatment and had data to report.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 4
units on a scale | 23.54 (12.80) | 37.75 (8.66)

2. Primary Outcome: Client Satisfaction Questionnaire-8
Description: Client Satisfaction Questionnaire-8 is a reliable and valid self-report of participants' acceptability of treatment. This is an assessment of client/patient satisfaction with their care and perceived quality and tolerability of NEW Tx. The scale for this item is a 4-point Likert scale ranging from 1 ("poor") to 4 ("excellent"). The score for each item is summed for a total score that ranges from 8 to 32 with higher scores indicating greater acceptability of the treatment.TAU participants only received this questionnaire if they chose to participate in the NEW Tx at week 20 of the intervention following the waitlist period.
Time Frame: 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
units on a scale | 25.77 (6.88) | 23.13 (8.11)

3. Secondary Outcome: LIFE- Range of Impaired Functioning Tool
Description: LIFE- Range of Impaired Functioning Tool assesses the extent to which medical burden has impacted current functioning. The score for each domain is summed for a total score that ranges from 4 to 20 with higher scores indicating worse functioning.
Time Frame: 20 weeks
Population: Results reported here include scores for participants at the post-treatment visit. Thus, these results only include data from participants who did not drop out by week 20 and had data to report.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 12
units on a scale | 9.08 (3.77) | 9.75 (3.33)

4. Secondary Outcome: Montgomery Asberg Depression Rating Scale
Description: Montgomery Asberg Depression Rating Scale is a 10-item clinician-rated measure of depression that assesses the presence and severity of patient's current depressive symptoms. The score for each item is summed for a total score that ranges from 0 to 60 with higher scores indicating more severe current depressive symptoms.
Time Frame: 20 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 12
units on a scale | 13.11 (8.89) | 12.36 (9.23)

5. Secondary Outcome: Young Mania Rating Scale
Description: Young Mania Rating Scale is an 11-item, clinician-rated measure that assesses the presence and severity of patient's current symptoms of mania. The score for each item is summed for a total score that ranges from 0 to 56 with higher scores indicating more severe current manic symptoms.
Time Frame: 20 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 12
units on a scale | 5.42 (8.55) | 5.95 (5.90)

6. Secondary Outcome: Body Mass Index (BMI)
Description: Body Mass Index levels at post-treatment.
Time Frame: 20 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11
kg/m^2 | 32.49 (4.29) | 35.76 (7.51)

7. Secondary Outcome: Weekly Exercise Duration
Description: Weekly exercise duration reported at post-treatment.
Time Frame: 20 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NEW Tx | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 12
minutes | 268.08 (242.72) | 85.42 (69.53)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | NEW Tx | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 5/19 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NEW Tx (N=19) | Treatment as Usual (TAU) (N=19)
Medical Issues (Physical) (Surgical and medical procedures) | 5 (5) | 2 (3) — Breaks, sprains, infection
Unrelated Life Events (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) — Life events unrelated to study procedures (e.g., car accident, work injury)
Worsening Psychiatric Illness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT01615367/Prot_SAP_000.pdf